CLINICAL TRIAL: NCT02335437
Title: Chronic Fatigue Following Acute Epstein-Barr Virus Infection in Adolescents
Acronym: CEBA
Status: Completed | Type: Observational
Sponsor: University Hospital, Akershus (Other)
Responsible Party: Principal Investigator, Vegard Bruun Wyller, MD, PhD, Professor, University Hospital, Akershus
Other Study IDs: CEBA
Record Dates: First submitted 2015-01-07; First posted 2015-01-09 (Estimated); Last update posted 2017-06-28 (Actual); Status verified 2017-06

CONDITIONS: Fatigue Syndrome, Chronic; Epstein-Barr Virus Infections
MeSH Terms: conditions — Fatigue Syndrome, Chronic; Epstein-Barr Virus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Acute EBV infection
- Healthy controls

SUMMARY:
Chronic fatigue syndrome (CFS) is characterized by unexplained, disabling and long lasting fatigue, as well as pain, impaired memory, sleep difficulties and other symptoms. Epstein-Barr virus (EBV) infection might precipitate CFS. In this study, 200 adolescents undergoing acute EBV infection will be followed prospectively, and also compared with a group of healthy controls. The aim is twofold:

* To identify factors that predispose to chronic fatigue among adolescents with acute EBV infection
* To compare pathophysiological features of patients with acute EBV infection with a group of healthy controls.

Possible risk factors for chronic fatigue 6 months after EBV-infection includes:

* Severity of the initial infection
* Immune responses characteristics
* Characteristics of the neuroendocrine stress response
* Cognitive functioning
* Emotional disturbances
* Genetics/ epigenetics of candidate genes
* Certain personality traits
* Critical life events

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 12 years and < 20 years
* Serological confirmation of acute EBV infection
* Lives in one of the following Norwegian counties: Oslo, Akershus, Buskerud, Østfold, Vestfold

Exclusion Criteria:

* Medical treatment for another disease (hormonal conterception and antibiotics against tonsillitis/pharyngitis are accepted)
* Pregnancy
* Debut of illness > 6 weeks ago

Ages: 12 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Microbiological laboratories serving the population of Oslo and neighbour conties.
Sampling Method: Probability Sample
Enrollment: 270 (Estimated)
Dates: Start 2015-03 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Fatigue | 6 monhts
  Chalder fatigue questionnaire, total score
Steps per day | 6 monhts
  Mean number of steps/day across 7 consecutive days, measured by accelerometer (ActivePal)

SECONDARY OUTCOMES:
Pain threshold | 6 monhts
  Assessed by pressure algometry
Autonomic cardiovascular control | 6 monhts
  Assessed by noninvasive, continuous recordings of heart rate, blood pressures and stroke volume during supine rest.
Cognitive function | 6 monhts
  Assessed by the instruments WISC-IV, D-KEFS, HVLT-R and WASI.
Neuroendocrine markers | 6 monhts
  In particular blood and urine measurements of catecholamines and the HPA axis
Immune markers | 6 monhts
  In particular blood measurements of cytokines
Bodily symptoms | 6 monhts
  Assessed by different questionnaires
Quality of life | 6 monhts
  Assessed by the PedsQL inventory
Functional disability | 6 monhts
  Assessed by the FDI inventory

CONTACTS AND LOCATIONS:
Overall Officials: Vegard B Wyller, Principal Investigator — University Hospital, Akershus
Locations (1):
- Dept. of Pediatrics, Akershus University Hospital, Lørenskog, Akershus, Norway

REFERENCES:
- [Derived] Fevang B, Wyller VBB, Mollnes TE, Pedersen M, Asprusten TT, Michelsen A, Ueland T, Otterdal K. Lasting Immunological Imprint of Primary Epstein-Barr Virus Infection With Associations to Chronic Low-Grade Inflammation and Fatigue. Front Immunol. 2021 Dec 20;12:715102. doi: 10.3389/fimmu.2021.715102. eCollection 2021. PMID 34987499
- [Derived] Pedersen M, Asprusten TT, Godang K, Leegaard TM, Osnes LT, Skovlund E, Tjade T, Oie MG, Wyller VBB. Predictors of chronic fatigue in adolescents six months after acute Epstein-Barr virus infection: A prospective cohort study. Brain Behav Immun. 2019 Jan;75:94-100. doi: 10.1016/j.bbi.2018.09.023. Epub 2018 Sep 25. PMID 30261303